CLINICAL TRIAL: NCT05428293
Title: Study of no Pharmacokinetic Interaction Between Ibuprofen 100 mg and Acetaminophen 125 mg, Suspension Administered Individually or in Combination, Single Dose in Healthy Subjects, Both Genders Under Fasting Conditions
Brief Title: Pharmacokinetic Interaction Between Ibuprofen and Acetaminophen Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BD IP-Sil No. 102-18
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Bioavailability; Fixed-dose combination (FDC); Ibuprofen; Acetaminophen; Oral suspension; Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Ibuprofen/ Acetaminophen oral suspension in fixed dose (Experimental): Pharmaceutical Form: Oral Suspension Formula: Ibuprofen 100 mg/ Acetaminophen 125 mg/ 5 mL Dosage: 5 mL Administration way: oral
  Interventions: Drug: A1: Ibuprofen/Acetaminophen Fixed dose combination oral suspension (Laboratorios Silanes S.A. de C.V.)
- Group B: Ibuprofen oral suspension (Active Comparator): Pharmaceutical Form: Oral Suspension Formula: Ibuprofen 2 g/100 mL Dosage: 5 mL (100 mg of ibuprofen) Administration way: oral
  Interventions: Drug: A2: Ibuprofen (Advil®, Pfizer S.A. de C.V.)
- Group C: Acetaminophen oral suspension (Active Comparator): Pharmaceutical Form: Oral Suspension Formula: Acetaminophen 3.2 g/100 mL Dosage: 3.9 mL (125 mg of acetaminophen) Administration way: oral
  Interventions: Drug: A3: Acetaminophen (Tylenol®, from Janssen-Cilag, S.A. de C.V.)

INTERVENTIONS:
Drug: A1: Ibuprofen/Acetaminophen Fixed dose combination oral suspension (Laboratorios Silanes S.A. de C.V.) — Formula : 100 mg/ 125 mg /5mL Pharmaceutical Form: Oral suspension Dosage: 5mL (100 mg/125mg) Administration way: oral
  Other Names: IBU/ACETA SUSP
  Arms: Group A: Ibuprofen/ Acetaminophen oral suspension in fixed dose
Drug: A2: Ibuprofen (Advil®, Pfizer S.A. de C.V.) — Pharmaceutical Form: oral suspension Formula: 2 g/100 mL Dosage: 5 mL(100 mg of Ibuprofen) Administration way: oral
  Other Names: IBU SUSP
  Arms: Group B: Ibuprofen oral suspension
Drug: A3: Acetaminophen (Tylenol®, from Janssen-Cilag, S.A. de C.V.) — Pharmaceutical Form: oral suspension Formula: 3.2 g/100 mL Dosage: 3.9 mL (125 mg) Administration way: oral
  Other Names: ACETA SUSP
  Arms: Group C: Acetaminophen oral suspension

SUMMARY:
This study was carried out in the Clinical and Analytical Unit of the Pharmacology and Toxicology Department of the Faculty of Medicine of the Autonomous University of Nuevo León, in order to compare the bioavailability (Cmax, AUC) of an oral formulation containing Ibuprofen 100 mg/Acetaminophen 125 mg in combination with the two oral formulations Ibuprofen 100 mg or Acetaminophen 125 mg administered as a single dose, in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
The study design was crossover, 3 x 6 x 3, open, prospective and longitudinal, at a single dose, of the combination of Ibuprofen 100 mg/Acetaminophen 125 mg/5 mL suspension, administered orally versus each component administered individually Ibuprofen 100 mg/5 mL or Acetaminophen 125 mg/3.9 mL, with an elimitation period (washout) of 1 week. In order to compare the pharmacokinetic profile (Cmax and AUC0-t) of the Ibuprofen/Acetaminophen combination 100 mg/125 mg/5 mL, versus each component administered individually, in 42 healthy subjects, of both genders, under fasting conditions, to establish the interaction of drugs in combination. As well as, to characterize the pharmacokinetic parameters, Cmax and AUC0-t, AUC0-∞, Tmax, Ke, and T1/2 and to establish the frequency and type of adverse events with the two formulations.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have been accepted by the COFEPRIS research subjects registration database.
* Subjects without a subordinate relationship with the researchers.
* Subjects who have given informed consent in writing.
* Subjects of both genders, aged between 18 and 55 years, Mexicans. - -Subjects with no background of hypersensitivity or allergies to the drug under study or related drugs.
* Body mass index between 18 and 27 kg/m2.
* Healthy subjects, according to the results of the complete clinical history, electrocardiogram and the integration of the results of the clinical analyses, carried out in certified clinical laboratories, without alterations that require a medical intervention as a consequence.
* Subjects with negative results for immunological tests (Anti-HIV, Anti-hepatitis B and C, VDRL).
* Subjects with negative results in drug abuse screening tests: tetrahydrocannabinoids, cocaine and amphetamines.
* Negative (qualitative) pregnancy test for women of childbearing potential without Bilateral tubal obstruction or hysterectomy.
* In the case of women of childbearing age, they must have a birth control method, including barrier methods, non-hormonal intrauterine device, or bilateral tubal obstruction.

Exclusion Criteria:

* Subjects with recent history or physical examination evidence of gastrointestinal, renal, hepatic, endocrine, respiratory, cardiovascular, dermatological, or hematological disease that could affect the pharmacokinetic study of the product in research.
* Subjects who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken drugs potentially toxic within 30 days before the start of the study.
* Subjects who have received any medication during the 7 days before the start of the study.
* Subjects who have been hospitalized for any problem during the three months before the start of the study.
* Subjects who have been rejected by the registry database of research subjects of COFEPRIS, for having participated in a clinical study within the three months prior to the start of the study.
* Subjects who have received investigational drugs within the previous 60 days th the start of the study.
* Subjects allergic to the study drug or related drugs.
* Subjects who have ingested alcohol or drinks containing xanthines (coffee, tea, cocoa, chocolate, cola) or who have eaten charcoal-grilled food or grapefruit juice , at least 10 hours before the start of the study or who have smoked tobacco 24 hours before to the start of the internment period.
* Subjects who have donated or lost 450 mL or more of blood within the previous 60 days of the beginning of the study. - Subjects with a history of drug and/or alcohol abuse according to the DSM-IV-TR Criteria.
* Research subjects who presents alterations in the vital signs recorded during the selection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose Ibuprofen/Acetaminophen oral suspension, employing the maximum observed concentration following the treatment (Cmax), obtained graphically, from the plasma concentration profile with respect to time.
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Ibuprofen/Acetaminophen oral suspension, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t) using the linear trapezoidal method.

SECONDARY OUTCOMES:
The area under the curve from time zero to infinity calculated (AUC 0-inf) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of ibuprofen/Acetaminophen oral suspension, employing the area under the curve from time zero to infinity calculated (AUC 0-inf)
Time of the maximum measured concentration (Tmax) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of ibuprofen/Acetaminophen oral suspension, employing time of the maximum measured concentration Tmax), obtained graphically, from the plasma concentration profile with respect to time.
Elimination rate (Ke) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of ibuprofen/Acetaminophen oral suspension, employing the elimination rate (Ke), estimated from the terminal linear portion of the plasma concentration profile with respect to time (on a semi-log scale)
Half time elimination (T1/2) | Baseline, 0.16, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12,0 and 14.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose ibuprofen/Acetaminophen oral suspension, employing the half time elimination (T1/2) by the quotient of Ln(2)Ke.
Frequency of occurrence of adverse events | 1, 8 and 16 days
  The percentage of frequency of appearance of each adverse event was evaluated.
Adverse events | 1, 8 and 16 days
  Any adverse event was classified by severity, treatment and its relationship with the study drug evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocaña, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Tanner T, Aspley S, Munn A, Thomas T. The pharmacokinetic profile of a novel fixed-dose combination tablet of ibuprofen and paracetamol. BMC Clin Pharmacol. 2010 Jul 5;10:10. doi: 10.1186/1472-6904-10-10. PMID 20602760
- [Background] Zhang Y, Mehrotra N, Budha NR, Christensen ML, Meibohm B. A tandem mass spectrometry assay for the simultaneous determination of acetaminophen, caffeine, phenytoin, ranitidine, and theophylline in small volume pediatric plasma specimens. Clin Chim Acta. 2008 Dec;398(1-2):105-12. doi: 10.1016/j.cca.2008.08.023. Epub 2008 Sep 3. PMID 18796299
- See also: Drugbank. Ibuprofen — https://www.drugbank.ca/atc/MO1AE01
- See also: Drugbank. Acetaminophen — https://www.drugbank.ca/atc/NO2BE01